CLINICAL TRIAL: NCT02402543
Title: Pre-Emptive Analgesia in Ano-Rectal Surgery
Acronym: PEAARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: American Society of Colon and Rectal Surgeons (Other)
Responsible Party: Principal Investigator, Peter Cataldo, MD, Professor of Surgery and Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHRMS: M13-226
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Hemorrhoids; Fissure in Ano; Rectal Fistula; Anal Condyloma
Keywords: preemptive analgesia; anorectal surgery; gabapentin; neurontin; ketamine; acetaminophen; tylenol; postoperative pain; postoperative narcotic usage; dexamethasone; decadron
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano; Rectal Fistula; Pain, Postoperative | interventions — Gabapentin; Ketamine; Acetaminophen; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Placebo Comparator): In pre-op, the subject is administered four placebo pills PO containing confectioners sugar, which are matched in color, size, and shape to the active pills.
  Interventions: Drug: Placebo
- Experimental Arm (Experimental): In pre-op, the subject is administered four pills PO containing a total of 1000 mg of acetaminophen and 600 mg of gabapentin, which are matched in color, size, and shape to the placebo pills.
  Interventions: Drug: Gabapentin; Drug: Ketamine; Drug: Acetaminophen; Drug: Dexamethasone

INTERVENTIONS:
Drug: Gabapentin
  Other Names: Neurontin, Gralise, Fanatrex
  Arms: Experimental Arm
Drug: Ketamine — Prior to the incision in the operating room, the anesthesiologist administers 0.15 mg/kg of ketamine IV push in patients randomized to the experimental arm, only.
  Other Names: Ketalar
  Arms: Experimental Arm
Drug: Acetaminophen
  Other Names: Tylenol, panadol, mapap, ofirmev, tempra
  Arms: Experimental Arm
Drug: Dexamethasone — Prior to the incision in the operating room, the anesthesiologist administers 8 mg of dexamethasone IV push in patients randomized to the experimental arm, only.
  Other Names: Decadron,
  Arms: Experimental Arm
Drug: Placebo
  Arms: Control Arm

SUMMARY:
The perianal region is the region around the anus. Administering a pain medication before a surgery starts is called preemptive analgesia. In some studies, this technique has been shown to be an effective way to reduce the pain that a patient experiences in the post-operative timeframe to a greater extent than would be expected simply from the pain medications alone. One theory of why this occurs suggests that the preemptive analgesia desensitizes brain and nerves to pain, thereby decreasing the response to painful stimuli, like surgery when they occur. This leads to a decrease in the amount of narcotic pain medication required after the procedure, which leads to less side effects and a quicker return to normal functioning. As perianal surgeries do not usually include a long stay in the hospital, controlling post-procedure pain is a priority.

The use of preemptive analgesia is in other types of surgeries, such as orthopedics, is well established, but as the perianal region has not been well studied, its use is not the standard of care. This type of analgesia uses a combination of medications that are already in use for post-operative and non-operative pain control and administers them orally prior to the patient undergoing general anesthesia. The side effects of the medications are the same as if they had been given after surgery or for non-surgical pain.

The concept of preemptive analgesia is established in other types of surgeries and it has solid basic science to support its use. The purpose of this randomized, double-blind, placebo controlled study is to determine if patients undergoing perianal surgeries could benefit from preemptive pain control. The primary outcome will be whether patients experience less post-operative pain. Patient post-operative consumption and latency until use of narcotic pain medication will be the secondary outcomes. The investigators believe that the patients receiving pain medications before their operation will require less pain medication after surgery, with minimal increased risk to the patient.

DETAILED DESCRIPTION:
Despite advances in pain medicine, postoperative pain control remains problematic with over 5% of patients experiencing severe pain despite standard of care pain management, and is a frequently cited reason for delayed discharge in outpatient procedures [1]. In anorectal surgeries, almost all patients experience mild-to-moderate postoperative subjective pain [2], and as an example 12% of patients report severe postoperative pain during their recovery from hemorrhoidectomy surgery [3]. Control of postoperative pain is an important goal. Preemptive analgesia is a technique that involves premedicating the patient with a regimen of medications designed to target different points in the pain cascade to prevent central and peripheral sensitization to pain, also known as "wind-up" [4]. The activation of N-methyl-D-aspartate (NMDA) receptors is an identified process that occurs in central sensitization after a noxious stimulus. By pharmacologically blocking these receptors, it may be possible to prevent or suppress the degree of central sensitization, which can prevent the hyperalgesic, or exaggerated pain response, that some patients experience [5]. Peripheral sensitization is a similar concept and occurs due to noxious stimuli in the periphery, such as a surgical incision. This type of sensitization has typically been prevented with regional anesthesia and by increasing the nociceptive threshold of the neurons with different medications.

Preemptive analgesia focusing on the effect of single medications on pain control has shown promising results, however some studies appear to lend themselves to practice [6-19] better than others [20-26]. On the other hand, multimodal pain control regimens might be more promising. A search of the literature reveals that preemptive pharmacological blockade of wind up has been effectively used in both surgical and nonsurgical patients (burn patients [27]). In patients undergoing hip arthroplasty, or hip replacement surgery, under general anesthesia, blocking both central and peripheral sensitization results in significantly decreased subjective pain, and a trend toward less postoperative use of analgesics [28]. Similarly, patients undergoing multilevel spinal surgeries [29] and those undergoing prostatic surgery [30] under general anesthesia consume less postoperative analgesics when undergoing multimodal preemptive pain control by blocking both sensitization pathways. Finally, preemptive central sensitization blockade alone has been used with trends in improved pain control for gynecological surgeries under both general [31] and regional anesthesia [32]. The preemptive use of such medications has not been studied for anorectal surgeries and it is what we are suggesting in this study. Most pain control studies in the literature focus on postoperative rather than preemptive medication regimens for pain management [33-35], and there is no current standard of care as to an effective regimen. The studies effective in decreasing postoperative pain in other surgical contexts, such as for patients undergoing hip arthroplasty, have used the same combination of medications proposed for the Treatment Group. Finally, the added benefit of the anorectal patient population in terms of the putative decreased use of opioids for postoperative pain control revolves around the opioid-related adverse effects on bowel function. In fact, return of bowel movements and regularity is one criterion for healing after surgery.

Based on this existing literature, we propose in our current study to preemptively block both central sensitization through the use of intravenous ketamine perioperatively and peripheral sensitization through the use of intravenous dexamethasone administered perioperatively and oral gabapentin and acetaminophen administered preoperatively. Ketamine is a noncompetitive NMDA receptor antagonist acting centrally in the dorsal horn of the spinal cord to decrease the release of glutamate, reducing the transmission of pain messages centrally [36]. Intravenous ketamine has been shown to decrease 24-hour opioid requirements, and preemptive use of ketamine was part of the medications used in most of the studies mentioned in the literature review above. As it currently stands, use of ketamine in anorectal surgeries as an added analgesic has been proven safe. Among Nigerian surgery patients having received regional anesthesia and preemptive ketamine, postoperative pain levels have been shown to decrease, however it is unclear if this patient cohort included anorectal surgery patients [37]. No other studies have been conducted regarding postoperative pain in these patients [38]. By utilizing ketamine as one of the medications in our study, we hope to show similar effects resulting in patients experiencing decreased postoperative pain after common anorectal surgeries.

Dexamethasone is a corticosteroid with potent anti-inflammatory effects that is also used as an anti-emetic. The proposed mechanism of action of dexamethasone is not completely known, but it is thought to involve inhibition of prostaglandin synthesis and an increased release of endorphins. Endorphins are endogenous peptides that bind to pain receptors in the body to decrease pain. In addition, endorphins can facilitate mood elevation and a sense of well-being. Intravenous dexamethasone was part of the medications used in studies mentioned in the literature review above. One study investigating the prophylactic use of dexamethasone for its anti-emetic properties, in combination with sevoflurane, a general anesthetic, during anorectal surgery found a significant decrease in maximal postoperative VAS pain scores in patients administered dexamethasone compared to those given placebos [2]. The use of dexamethasone as a preemptive analgesic has not been fully studied in anorectal surgery patients.

Gabapentin acts by binding to receptors on voltage-gated calcium channels on presynaptic nerves, reducing the entry of calcium into presynaptic nerve terminals. The subsequent decreased release of excitatory neurotransmitters such as glutamate, aspartate, substance P, and norepinephrine into the synaptic cleft is linked to a diminished postsynaptic transmission of neural pain messages [36]. It is usually used for neuropathic pain control, and has been used in some of the studies mentioned in the literature review above. A systemic review of the perioperative effects of gabapentin found that it is an effective means of reducing post-operative pain, opioid consumption, and opioid-related adverse effects in surgical patients. In fact, administration of a single dose of gabapentin was found to be equivalent to a reduction of 30 mg of morphine in the first 24 hours after surgery [39]. No studies have been conducted, to the best of our knowledge, regarding preemptive use of gabapentin in anorectal surgeries.

Local, peripheral sensitization has also been minimized through the use of non-steroidal anti-inflammatory drugs (NSAIDs) due to the decreased production of certain molecules such as prostaglandins and kinins. The enzyme required to make these molecules is blocked by acetaminophen and NSAIDs, which is why acetaminophen is included in this study in hopes of demonstrating better pain control among anorectal surgery patients. Acetaminophen is a weak analgesic that forms the most basic component of a multimodal analgesia regimen [36]. Oral preemptive use of acetaminophen has been proven to decrease postoperative narcotic use in surgical patients [40], and has been used in some of the studies mentioned in the literature review above. A related intramuscular NSAID, namely Toradol, has been used preemptively among anorectal surgical patients with good pain control [41]. No other studies are reported in this patient population.

Of importance, the combinations of the medications used in this study have been used in other studies before with similar or higher doses and no significant differences in terms of hemodynamic variables (such as vital signs) or adverse side effects have been noted compared to control groups [31]. In fact, these medications are safely used at UVM Medical Center by the collaborating surgeons as part of their care for other surgeries such as abdominal surgeries.

*References 1-41 available upon request

ELIGIBILITY:
Inclusion Criteria:

* Patients having anal fistula repairs for anal fistulas recalcitrant to non-surgical management at the University of Vermont Medical Center or Fanny Allen Campuses OR
* Patients having anal sphincterotomies for chronic anal fissures recalcitrant to non-surgical management at the University of Vermont Medical Center or Fanny Allen Campuses OR
* Patients having hemorrhoidectomies for hemorrhoids recalcitrant to non-surgical management at the University of Vermont Medical Center or Fanny Allen Campuses OR
* Patients having anal condyloma excisions for anal condylomas recalcitrant to non-surgical management at the University of Vermont Medical Center or Fanny Allen Campuses
* Patients undergoing these surgeries must be American Society of Anesthesiologists (ASA) Physical Status Classification System scores of I (normal, healthy patient), II (patient with mild, systemic disease), or III (patients with more significant disease)

Exclusion Criteria:

* Allergies to any study medications;
* Patient history and chart review for existence of hepatic or renal failure;
* Chronic pain syndrome;
* Inability to understand or utilize the Numerical Rating Scale (NRS);
* Pregnancy;
* Patients currently on gabapentin, pregabalin or narcotics
* Patients taking chronic steroids, unable to taper off before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | End of surgery up to 7 days postoperatively
  Pain will be evaluated using numerical rating scales at specified intervals from the end of surgery up to 7 days postoperatively and mailed back to the investigators. The pain levels will be compared between groups.

SECONDARY OUTCOMES:
Narcotic consumption | End of surgery up to 7 days postoperatively
  Narcotic consumption will be recorded by the subject on medication diaries attached to the respective numerical rating scale. This helps to identify at which time point the patient took a narcotic. This will be compared between groups.
Interval for rescue pain medication | End of surgery up to 7 days postoperatively
  On the aforementioned medication diaries, the patient will record when he or she first needed break through pain medication (i.e. the narcotic prescribed) beyond the scheduled pain medicines. This will help us evaluate the interval between end of the operation and first need for breakthrough pain medication. This number will be compared between groups.
Further pain requirements | End of surgery up to 7 days postoperatively
  By examining the medication diaries, we will be able to evaluate if there were patients who required more than the scheduled pain medications and breakthrough narcotic. This number will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont Medical Center Fanny Allen Campus, Colchester, Vermont

REFERENCES:
- [Background] Chung F, Ritchie E, Su J. Postoperative pain in ambulatory surgery. Anesth Analg. 1997 Oct;85(4):808-16. doi: 10.1097/00000539-199710000-00017. PMID 9322460
- [Background] Wu JI, Lu SF, Chia YY, Yang LC, Fong WP, Tan PH. Sevoflurane with or without antiemetic prophylaxis of dexamethasone in spontaneously breathing patients undergoing outpatient anorectal surgery. J Clin Anesth. 2009 Nov;21(7):469-73. doi: 10.1016/j.jclinane.2008.11.007. PMID 19914051
- [Background] Labas P, Ohradka B, Cambal M, Olejnik J, Fillo J. Haemorrhoidectomy in outpatient practice. Eur J Surg. 2002;168(11):619-20. doi: 10.1080/11024150201680008. PMID 12699098
- [Background] MENDELL LM, WALL PD. RESPONSES OF SINGLE DORSAL CORD CELLS TO PERIPHERAL CUTANEOUS UNMYELINATED FIBRES. Nature. 1965 Apr 3;206:97-9. doi: 10.1038/206097a0. No abstract available. PMID 14334366
- [Background] Stubhaug A, Breivik H, Eide PK, Kreunen M, Foss A. Mapping of punctuate hyperalgesia around a surgical incision demonstrates that ketamine is a powerful suppressor of central sensitization to pain following surgery. Acta Anaesthesiol Scand. 1997 Oct;41(9):1124-32. doi: 10.1111/j.1399-6576.1997.tb04854.x. PMID 9366932
- [Background] Jirasiritham S, Tantivitayatan K, Jirasiritham S. Perianal blockage with 0.5% bupivacaine for postoperative pain relief in hemorrhoidectomy. J Med Assoc Thai. 2004 Jun;87(6):660-4. PMID 15279345
- [Background] Wnek W, Zajaczkowska R, Wordliczek J, Dobrogowski J, Korbut R. Influence of pre-operative ketoprofen administration (preemptive analgesia) on analgesic requirement and the level of prostaglandins in the early postoperative period. Pol J Pharmacol. 2004 Sep-Oct;56(5):547-52. PMID 15591642
- [Background] Lavand'homme P, De Kock M, Waterloos H. Intraoperative epidural analgesia combined with ketamine provides effective preventive analgesia in patients undergoing major digestive surgery. Anesthesiology. 2005 Oct;103(4):813-20. doi: 10.1097/00000542-200510000-00020. PMID 16192774
- [Background] Rockemann MG, Seeling W, Bischof C, Borstinghaus D, Steffen P, Georgieff M. Prophylactic use of epidural mepivacaine/morphine, systemic diclofenac, and metamizole reduces postoperative morphine consumption after major abdominal surgery. Anesthesiology. 1996 May;84(5):1027-34. doi: 10.1097/00000542-199605000-00003. PMID 8623995
- [Background] Kara I, Tuncer S, Erol A, Reisli R. [The effects of preemptive dexketoprofen use on postoperative pain relief and tramadol consumption]. Agri. 2011 Jan;23(1):18-21. doi: 10.5505/agri.2011.21939. Turkish. PMID 21341148
- [Background] Aida S, Yamakura T, Baba H, Taga K, Fukuda S, Shimoji K. Preemptive analgesia by intravenous low-dose ketamine and epidural morphine in gastrectomy: a randomized double-blind study. Anesthesiology. 2000 Jun;92(6):1624-30. doi: 10.1097/00000542-200006000-00020. PMID 10839912
- [Background] Zielinski J, Jaworski R, Smietanska I, Irga N, Wujtewicz M, Jaskiewicz J. A randomized, double-blind, placebo-controlled trial of preemptive analgesia with bupivacaine in patients undergoing mastectomy for carcinoma of the breast. Med Sci Monit. 2011 Oct;17(10):CR589-97. doi: 10.12659/msm.881986. PMID 21959614
- [Background] Kilickan L, Toker K. The effect of preemptive intravenous morphine on postoperative analgesia and surgical stress response. Panminerva Med. 2001 Sep;43(3):171-5. PMID 11579330
- [Background] Cai XH, Wang SP, Chen XT, Peng SL, Cao MH, Ye XJ, Yang YZ. [Comparison of three analgesic methods for postoperative pain relief and their effects on plasma interleukin-6 concentration following radical surgery for gastric carcinoma]. Nan Fang Yi Ke Da Xue Xue Bao. 2007 Mar;27(3):387-9. Chinese. PMID 17426001
- [Background] Ng WT. Re: laparoscopic repair of colonoscopic perforations. Surg laparosc endosc percutan tech. 2006;16:49-51. Surg Laparosc Endosc Percutan Tech. 2007 Feb;17(1):68-9; author reply 69. doi: 10.1097/01.sle.0000213751.23396.9e. No abstract available. PMID 17318064
- [Background] Wang Q, Li Z, Wang ZP, Cui C. [Preemptive analgesic effect of parecoxib sodium in patients undergoing laparoscopic colorectal surgery]. Nan Fang Yi Ke Da Xue Xue Bao. 2010 Nov;30(11):2556-7. Chinese. PMID 21097433
- [Background] Yeh CC, Jao SW, Huh BK, Wong CS, Yang CP, White WD, Wu CT. Preincisional dextromethorphan combined with thoracic epidural anesthesia and analgesia improves postoperative pain and bowel function in patients undergoing colonic surgery. Anesth Analg. 2005 May;100(5):1384-1389. doi: 10.1213/01.ANE.0000148687.51613.B5. PMID 15845691
- [Background] Fu ES, Miguel R, Scharf JE. Preemptive ketamine decreases postoperative narcotic requirements in patients undergoing abdominal surgery. Anesth Analg. 1997 May;84(5):1086-90. doi: 10.1097/00000539-199705000-00024. PMID 9141936
- [Background] Clarke H, Pereira S, Kennedy D, Andrion J, Mitsakakis N, Gollish J, Katz J, Kay J. Adding gabapentin to a multimodal regimen does not reduce acute pain, opioid consumption or chronic pain after total hip arthroplasty. Acta Anaesthesiol Scand. 2009 Sep;53(8):1073-83. doi: 10.1111/j.1399-6576.2009.02039.x. Epub 2009 Jun 30. PMID 19572933
- [Background] Abramov Y, Sand PK, Gandhi S, Botros SM, Miller JJ, Koh EK, Goldberg RP. The effect of preemptive pudendal nerve blockade on pain after transvaginal pelvic reconstructive surgery. Obstet Gynecol. 2005 Oct;106(4):782-8. doi: 10.1097/01.AOG.0000165275.39905.0d. PMID 16199636
- [Background] Fassoulaki A, Sarantopoulos C, Zotou M, Papoulia D. Preemptive opioid analgesia does not influence pain after abdominal hysterectomy. Can J Anaesth. 1995 Feb;42(2):109-13. doi: 10.1007/BF03028261. PMID 7720151
- [Background] Holthusen H, Backhaus P, Boeminghaus F, Breulmann M, Lipfert P. Preemptive analgesia: no relevant advantage of preoperative compared with postoperative intravenous administration of morphine, ketamine, and clonidine in patients undergoing transperitoneal tumor nephrectomy. Reg Anesth Pain Med. 2002 May-Jun;27(3):249-53. doi: 10.1053/rapm.2002.30669. PMID 12016597
- [Background] Romej M, Voepel-Lewis T, Merkel SI, Reynolds PI, Quinn P. Effect of preemptive acetaminophen on postoperative pain scores and oral fluid intake in pediatric tonsillectomy patients. AANA J. 1996 Dec;64(6):535-40. PMID 9204788
- [Background] Radhakrishnan M, Bithal PK, Chaturvedi A. Effect of preemptive gabapentin on postoperative pain relief and morphine consumption following lumbar laminectomy and discectomy: a randomized, double-blinded, placebo-controlled study. J Neurosurg Anesthesiol. 2005 Jul;17(3):125-8. doi: 10.1097/01.ana.0000167147.90544.ab. PMID 16037731
- [Background] Canbay O, Karakas O, Celebi N, Peker L, Coskun F, Aypar U. The preemptive use of diclofenac sodium in combination with ketamine and remifentanil does not enhance postoperative analgesia after laparoscopic gynecological procedures. Saudi Med J. 2006 May;27(5):642-5. PMID 16680253
- [Background] Richardson P, Mustard L. The management of pain in the burns unit. Burns. 2009 Nov;35(7):921-36. doi: 10.1016/j.burns.2009.03.003. Epub 2009 Jun 7. PMID 19505764
- [Background] Rasmussen ML, Mathiesen O, Dierking G, Christensen BV, Hilsted KL, Larsen TK, Dahl JB. Multimodal analgesia with gabapentin, ketamine and dexamethasone in combination with paracetamol and ketorolac after hip arthroplasty: a preliminary study. Eur J Anaesthesiol. 2010 Apr;27(4):324-30. doi: 10.1097/EJA.0b013e328331c71d. PMID 19734790
- [Background] Mathiesen O, Dahl B, Thomsen BA, Kitter B, Sonne N, Dahl JB, Kehlet H. A comprehensive multimodal pain treatment reduces opioid consumption after multilevel spine surgery. Eur Spine J. 2013 Sep;22(9):2089-96. doi: 10.1007/s00586-013-2826-1. Epub 2013 May 17. PMID 23681498
- [Background] Trabulsi EJ, Patel J, Viscusi ER, Gomella LG, Lallas CD. Preemptive multimodal pain regimen reduces opioid analgesia for patients undergoing robotic-assisted laparoscopic radical prostatectomy. Urology. 2010 Nov;76(5):1122-4. doi: 10.1016/j.urology.2010.03.052. Epub 2010 Jun 8. PMID 20570321
- [Background] Kwok RFK, Lim J, Chan MTV, Gin T, Chiu WKY. Preoperative ketamine improves postoperative analgesia after gynecologic laparoscopic surgery. Anesth Analg. 2004 Apr;98(4):1044-1049. doi: 10.1213/01.ANE.0000105911.66089.59. PMID 15041596
- [Background] Menkiti ID, Desalu I, Kushimo OT. Low-dose intravenous ketamine improves postoperative analgesia after caesarean delivery with spinal bupivacaine in African parturients. Int J Obstet Anesth. 2012 Jul;21(3):217-21. doi: 10.1016/j.ijoa.2012.04.004. Epub 2012 Jun 1. PMID 22658477
- [Background] Luck AJ, Hewett PJ. Ischiorectal fossa block decreases posthemorrhoidectomy pain: randomized, prospective, double-blind clinical trial. Dis Colon Rectum. 2000 Feb;43(2):142-5. doi: 10.1007/BF02236970. PMID 10696885
- [Background] Vinson-Bonnet B, Coltat JC, Fingerhut A, Bonnet F. Local infiltration with ropivacaine improves immediate postoperative pain control after hemorrhoidal surgery. Dis Colon Rectum. 2002 Jan;45(1):104-8. doi: 10.1007/s10350-004-6121-4. PMID 11786772
- [Background] Tegon G, Pulzato L, Passarella L, Guidolin D, Zusso M, Giusti P. Randomized placebo-controlled trial on local applications of opioids after hemorrhoidectomy. Tech Coloproctol. 2009 Sep;13(3):219-24. doi: 10.1007/s10151-009-0518-y. Epub 2009 Aug 1. PMID 19649687
- [Background] Tang R, Evans H, Chaput A, Kim C. Multimodal analgesia for hip arthroplasty. Orthop Clin North Am. 2009 Jul;40(3):377-87. doi: 10.1016/j.ocl.2009.04.001. PMID 19576406
- [Background] Famewo CE. Study of incidence of post-operative pain among Nigerian patients. Afr J Med Med Sci. 1985 Sep-Dec;14(3-4):175-9. PMID 3004177
- [Background] Sun MY, Canete JJ, Friel JC, McDade J, Singla S, Paterson CA, Counihan TC. Combination propofol/ketamine is a safe and efficient anesthetic approach to anorectal surgery. Dis Colon Rectum. 2006 Jul;49(7):1059-65. doi: 10.1007/s10350-006-0572-8. PMID 16699969
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Background] Khalili G, Janghorbani M, Saryazdi H, Emaminejad A. Effect of preemptive and preventive acetaminophen on postoperative pain score: a randomized, double-blind trial of patients undergoing lower extremity surgery. J Clin Anesth. 2013 May;25(3):188-92. doi: 10.1016/j.jclinane.2012.09.004. Epub 2013 Apr 6. PMID 23567482
- [Background] Richman IM. Use of Toradol in anorectal surgery. Dis Colon Rectum. 1993 Mar;36(3):295-6. doi: 10.1007/BF02053515. PMID 8449138
- [Background] Poylin V, Quinn J, Messer K, Nagle D. Gabapentin significantly decreases posthemorrhoidectomy pain: a prospective study. Int J Colorectal Dis. 2014 Dec;29(12):1565-9. doi: 10.1007/s00384-014-2018-4. Epub 2014 Oct 1. PMID 25269619